CLINICAL TRIAL: NCT05549258
Title: An Open-Label Multicenter Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Safety of Inebilizumab in Pediatric Subjects With Neuromyelitis Optica Spectrum Disorder
Brief Title: Study of Inebilizumab in Pediatric Subjects With Neuromyelitis Optica Spectrum Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIB0551.P2.S2.NMO; 2023-510007-22 (EudraCT Number)
Expanded Access: NCT06590051 (Available)
Record Dates: First submitted 2022-07-22; First posted 2022-09-22 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Neuromyelitis Optica Spectrum Disorder
Keywords: NMOSD
MeSH Terms: conditions — Neuromyelitis Optica | interventions — inebilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Inebilizumab (Experimental): Infusion of Inebilizumab
  Interventions: Drug: Inebilizumab

INTERVENTIONS:
Drug: Inebilizumab — Inebilizumab administered intravenously (IV) over a total of 28 weeks.

SUMMARY:
A Phase 2, open-label, multicenter study to evaluate the pharmacokinetics (PK), pharmacodynamics (PD), and safety of inebilizumab in eligible pediatric participants 2 to < 18 years of age with recently active neuromyelitis optica spectrum disorder (NMOSD) who are seropositive for autoantibodies against aquaporin-4 (AQP4-immunoglobulin [Ig]G).

DETAILED DESCRIPTION:
Approximately 15 participants to be enrolled and receive Inebilizumab administered intravenously over 28 weeks. The maximum trial duration per participant is approximately 80 weeks, including up to 4 week screening period, 9 visits during a 28 week open-label treatment period, and approximately 4 visits during a 52 week follow-up period. Safety evaluations will be performed regularly throughout the course of the study.

Acquired from Horizon in 2023.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, minimum body weight of 15 kg, age 2 to < 18 years at the time of screening.
* Positive serum anti-AQP4-IgG result at screening and diagnosed with NMOSD according to the criteria of Wingerchuk et al, 2015.
* Documented history of one or more NMOSD acute relapses within the last year, or 2 or more NMOSD acute relapses within 2 years prior to screening.

Exclusion Criteria:

* Any condition that, in the opinion of the Investigator, would interfere with the evaluation or administration of the Investigational Product or interpretation of participant safety or study results.
* Concurrent/previous enrollment in another clinical study involving an investigational treatment within 4 weeks or 5 published half-lives of the investigational treatment, whichever is the longer, prior to Day 1.
* Evidence of significant hepatic, renal, or metabolic dysfunction or significant hematological abnormality (one repeat test may be conducted to confirm results within the same screening period).
* B-cell counts < one-half of the lower limit of normal (LLN) for age according to the central laboratory.
* Receipt of the following at any time prior to Day 1:

  1. Alemtuzumab
  2. Total lymphoid irradiation
  3. Bone marrow transplant
  4. T-cell vaccination therapy
* Receipt of rituximab or any experimental B-cell depleting agent within 6 months prior to screening unless B-cell counts have returned to ≥ one-half the LLN.
* Receipt of intravenous immunoglobulin (IVIG) within one month prior to Day 1.
* Receipt of any of the following within 2 months prior to Day 1:

  1. Cyclosporine
  2. Methotrexate
  3. Mitoxantrone
  4. Cyclophosphamide
  5. Tocilizumab
  6. Satralizumab
  7. Eculizumab
* Receipt of natalizumab (Tysabri®) within 6 months prior to Day 1.
* Severe drug allergic history or anaphylaxis to 2 or more food products or medicine (including known sensitivity to acetaminophen/paracetamol, diphenhydramine or equivalent antihistamine, and methylprednisolone or equivalent glucocorticoid).
* Diagnosed with a concurrent autoimmune disease that is uncontrolled (unless approved by the medical monitor).
* Recent receipt of live/attenuated vaccine or blood transfusion.

Receipt of any of the following:

1. Any live or attenuated vaccine within 4 weeks prior to Day 1 (administration of killed vaccines and nucleoside-modified mRNA-based vaccines is acceptable; the Sponsor recommends that Investigators ensure all participants are up to date on required vaccinations prior to study entry).
2. Bacillus Calmette Guérin vaccine within one year of screening.
3. Blood transfusion within 4 weeks prior to screening or during screening.

   * Clinically significant serious active or chronic viral, bacterial, or fungal infection that requires treatment with anti-infectives, hospitalization, or, in the Investigator's opinion, represents an additional risk to the participant, within 2 months prior to Day 1.
   * Known history of congenital or acquired immunodeficiency (e.g., due to human immunodeficiency virus [HIV] infection, splenectomy, immunosuppression-related or idiopathic T-cell deficiencies) that predisposes the participant to infection.
   * Positive test for chronic hepatitis B infection at screening, defined as either:

a. Positive hepatitis B surface antigen (HBsAg), or b. Positive hepatitis B core (HBc) antibody (anti-HBc) plus negative hepatitis B surface (HBs) antibody (anti-HBs).

* Positive test for hepatitis C virus antibody.
* Negative test for varicella zoster virus (VZV)-IgG.
* History of cancer, apart from squamous cell or basal cell carcinoma of the skin treated with documented success of curative therapy > 3 months prior to Day 1.
* History of active or latent tuberculosis (TB), or a positive QuantiFERON®-TB Gold test at screening, unless treatment for TB was completed per local guidelines. Participants with latent TB or a positive QuantiFERON®-TB Gold test who are actively on anti-TB treatment can enroll if they have completed at least one month of anti-TB treatment and intend to complete the full course of anti-TB treatment. Participants with an indeterminate QuantiFERON®-TB Gold test result can enroll if a repeat QuantiFERON®-TB Gold test is negative or a tuberculin skin test is negative.
* For participants who may undergo MRI scans:

  1. Unable to undergo an MRI scan (e.g., hypersensitivity to Gd-containing MRI contrast agents, implanted pacemakers, defibrillators, or other metallic objects on or inside the body that limit performing MRI scans), or
  2. Unable to tolerate or comply with the MRI procedure.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2027-04-13 (Estimated); Study Completion 2027-04-13 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) of Inebilizumab | Day 1 to Week 28
Area Under the Concentration Versus Time Curve of Inebilizumab from Time 0 to 14 Days Post-dose (AUC0-14d) | Day 1 to pre-dose on Day 15
Area Under the Concentration Versus Time Curve of Inebilizumab from Time 0 Extrapolated to Infinity (AUC0-Inf) | Day 1 to Week 80
Systemic Clearance (CL) of Inebilizumab | Day 1 to Week 80
Terminal Elimination Half-life (t½) of Inebilizumab | Day 1 to Week 80
Volume of Distribution at Steady State (VSS) of Inebilizumab | Day 1 to Week 80
Change from Baseline in Peripheral Cluster of Differentiation (CD)20-positive B-cell Counts | Week 1, Week 2, Week 28, Week 80
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Adverse Events of Special Interest (AESIs) | Day 1 to Week 80
Change from Baseline in Serum Chemistry | Week 1, Week 2, Week 28, Week 80
Change from Baseline in Hematology | Week 1, Week 2, Week 28, Week 80
Change from Baseline in Serum Immunoglobulins | Week 1, Week 2, Week 28, Week 80
Change from Baseline in Systolic Blood Pressure | Week 1, Week 2, Week 28, Week 80
Change from Baseline in Diastolic Blood Pressure | Week 1, Week 2, Week 28, Week 80
Change from Baseline in Pulse Rate | Week 1, Week 2, Week 28, Week 80
Change from Baseline in Respiratory Rate | Week 1, Week 2, Week 28, Week 80
Change from Baseline in Body Temperature | Week 1, Week 2, Week 28, Week 80

SECONDARY OUTCOMES:
Disease Activity: Time to First Relapse | Day 1 to Week 80
Disease Activity: Proportion of Relapse-free Participants | Day 1 to Week 80
Disease Activity: Annualized Relapse Rate | Day 1 to Week 80
Health-Related Quality of Life (HRQoL) change from baseline in Euro Quality of Life-5 Dimension Youth score | Day 1 to Week 80
  Change in baseline for the 5 dimensions: mobility, looking after myself, doing usual activities, having pain or discomfort, and feeling worried, sad, or unhappy. A higher score indicates onset or worsening of an affective disorder.
HRQoL change from baseline in Pediatric Quality of Life Inventory | Day 1 to Week 80
  Change in baseline comprised from 4 generic core scales: Physical Functioning, Emotional Functioning, Social Functioning, and School Functioning. A higher score indicates a better quality of life.
Visual Acuity change from baseline | Day 1 to Week 80
Change From Baseline in Expanded Disability Status Scale | Day 1 to Week 80
  Change in baseline comprised from results of 8 Functional Systems: Visual, Brainstem, Pryamidal, Cerebellar, Sensory, Bowel, Bladder, and Cerebral. A higher score indicates a higher grade of impairment and disability.
Anti-drug antibody (ADA) rate | Day 1 to Week 80

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (19):
- United States (4):
  - UCSD Altman Clinical and Translational Research Institute Building, La Jolla, California
  - Loma Linda University Children's Hospital - PIN, Loma Linda, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Hospital de Pediatría S.A.M.I.C.- Prof. Dr. Juan P. Garrahan, Parque Patricios, Ciudad Autónoma de BuenosAires, Argentina
- Brazil (4):
  - Hospital Santa Izabel-Rua Floriano Peixoto 300, Salvador, Estado de Bahia
  - Hospital Sao Lucas Da Pontificia Universidade Catolica Do Rio Grande Do Sul (PUCRS), Porto Alegre/RS
  - CPQuali Pesquisa Clínica Sao Paulo, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo
- Hospital For Sick Children, Toronto, Ontario, Canada
- Centre Hospitalier Universitaire de Bicêtre, Le Kremlin-Bicêtre, Val-de-Marne, France
- Erasmus MC Sophia Children's Hospital-Wytemaweg 80, Rotterdam, South Holland, Netherlands
- Uniwersyteckie Centrum Kliniczne w Gdansku - Smoluchowskiego 17, Gdansk, Poland
- Clinic for Neurology and Psychiatry for Children and Youth, Belgrade, Belgrade, Serbia
- Hospital Sant Joan de Deu - PIN, Espluges de Llobregat, Barcelona, Spain
- Karolinska Universitetssjukhuset Solna, Stockholm, Stockholm County, Sweden
- United Kingdom (3):
  - Evelina London Children's Hospital, London, London, City of
  - Great Ormond Street Hospital - PPDS, London, London, City of
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham, West Midlands

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com